CLINICAL TRIAL: NCT03162666
Title: Post-market Surveillance Study of Altera™ Minimally Invasive Articulating Expandable Spacer in a TLIF Interbody Fusion Device
Brief Title: Patient Outcomes Using an Expandable Spacer
Status: Withdrawn | Type: Observational
Why Stopped: The participating party (Rush) stopped the study because of logistic issues.
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RGC16-001
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2020-09

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ALTERA — degenerative disc disease (DDD) at one or two contiguous levels from L2 to S1. with up to grade 1 spondylolisthesis

SUMMARY:
This study is a post-market clinical follow-up study. The data collected from this study will serve the purpose of confirming safety and performance of the ALTERA™ Expandable implant.

DETAILED DESCRIPTION:
The evaluation is based on the following elements.

1. Safety as measured by the rate of serious operative and post-operative complications.
2. Subjects quality of life, measured by health-related quality of life questionnaires and Subject-reported outcome measures up to 24 months following the procedure, as compared to Subject's preoperative baseline.
3. Global and segmental lumbar lordosis (LL)

Patients will be followed upto 24 months post-operative

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-70 y/o)
* Male or Female
* With the following conditions of the lumbar spine as confirmed by advanced imaging (CT or MRI), who is a candidate for primary spinal fusion procedure according to acceptable criteria for such medical conditions:

  * Degenerative disc disease with up to Grade I spondylolisthesis
  * Spondylolisthesis
* Failure of at least 6-months conservative treatment
* BMI < 40
* Subject to approve no pregnancy during the 24 months of study and no participation in other studies in parallel to this one
* Ability to read, understand, and sign informed consent

Exclusion Criteria:

* Infection, local to the operative site
* Signs of local inflammation
* Fever or leukocytosis
* Pregnancy
* Significant mental disorder or condition that could compromise the Subject's ability to remember and comply with preoperative and postoperative instructions (e.g. current treatment for a psychiatric/psychosocial disorder, senile dementia, Alzheimer's disease, traumatic head injury)
* Prior surgical procedure (with the exception of decompression only procedure) at the index level(s) using the desired operative approach
* Prior fusion procedure at an adjacent level
* Any other condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumors or congenital abnormalities, fracture local to the operating site, elevation of segmentation rate unexplained by other diseases, elevation of white blood count (WBC), or a marked left shift in the WBC differential count
* Neuromuscular disorder that would engender unacceptable risk of instability, implant fixation failure, or complications in postoperative care
* Active local infection in or near the operative region
* Active systemic infection and/or disease
* Severe osteoporosis or insufficient bone density, which in the medical opinion of the physician precludes surgery or contraindicates instrumentation
* Endocrine or metabolic disorders known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, hypothyroidism)
* Systemic disease that requires the chronic administration of nonsteroidal anti-inflammatory or steroidal drugs
* Suspected or documented allergy or intolerance to implant's materials
* Symptomatic cardiac disease
* Subject unwilling to cooperate with postoperative instructions.
* Any case where the implant components selected for use would be too large or too small to achieve a successful result.
* Subject having inadequate tissue coverage over the operative site or inadequate bone stock or quality.
* Any Subject in which implant utilization would interfere with anatomical structures or expected physiological performance.
* Prior fusion at the level to be treated.
* Back VAS < 4/10

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that present to Rush University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2020-11-06 (Estimated); Study Completion 2020-11-06 (Estimated)

PRIMARY OUTCOMES:
Change in Radiographic Analysis | Pre-Op, 6weeks, 12 weeks, 6months, 12 months, 24 months
  Global and Segmental Lumbar Lordosis in degrees

SECONDARY OUTCOMES:
Complications | Intra-operative, any time post-op upto 24 months
  Surgical or device related complications
Change in Patient Reported Outcomes as a number score | Pre-Op, 6weeks, 12 weeks, 6months, 12 months, 24 months
  Visual Analog Scale, Oswestry Disability Index, Short Form 12, PROMIS
Peri operative clinical parameters | Intra-Operative
  Estimated Blood Loss in cc
Clinical parameters in days | Immediate Post-operative
  Length of Hospital Stay
Peri operative clinical parameters in mgs | Immediate Post-operative
  Narcotic Consumption
Intra-Operative clinical parameters in minutes | Intra-Operative
  Operative Time
Changes in Radiographic Analysis in percentage | 6weeks, 12 weeks, 6months, 12 months, 24 months
  Fusion Rates

CONTACTS AND LOCATIONS:
Overall Officials: Kern Singh, MD, Principal Investigator — Rush Univeristy Medical Center Orthopedic Surgeon
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No